CLINICAL TRIAL: NCT06922149
Title: Effects of Functional Massage Combined With Eccentric Exercise on Muscle Tone and Motor Function of the Lower Limb in Patients With Chronic Stroke: A Pilot Randomized Clinical Trial
Brief Title: Functional Massage and Eccentric Exercise in Stroke Survivors (FM-EE Stroke)
Acronym: FM-EE-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, Rosa Cabanas Valdés, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FM and EE stroke
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: stroke, eccentric exercises, functional massage, muscle tone
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A type of clinical trial in which all participants receive the same two treatments, but the order in which they receive them depends on the group to which they are randomly assigned. All participants will receive all the interventions but the order in which they will receive the interventions (the sequence) is randomised One group will get Group A during the first period of the trial, then Group B during the second period. A week of rest will be between groups.
  The other group will get Group B during the first period of the trial, then Group A during the second period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A Functional massage in addition to eccentric exercise in paretic lower limb (Experimental): Functional massage (FM) in addition to eccecntric exercises in paretic lower limb. FM is a massage technique that incorporates non-end-range joint motion (passive, active assisted or active) with massage (tissue compression) to treat musculotendinous dysfunction. During FM application, the target muscle and its surrounding soft tissues are compressed and the associated joint is moved to cause muscle lengthening or shortening. Shortening, or approximation, is used to aid the tissue in dispersing metabolic waste and improve the healing matrix of the injured tissue. Lengthening is used during the remodeling phase of tissue healing to improve mechanical strength, flexibility, and rigidity of the tissue. A combination of the two types can be used to aid in restoring the normal gliding of the connective tissue fibers during function. Eccentric resistance training is a method to improve strength and function that emphasizes the eccentric phase of the muscular contraction.
  Interventions: Other: Group A Funtional massage therapy and eccentric exercise in lower limb
- Group B Eccentric exercise in paretic lower limb (Active Comparator): Eccecntric exercises in paretic lower limb. Eccentric resistance training is a method to improve strength and function that emphasizes the eccentric phase of the muscular contraction. Some studies concluded that it allows the subject to produce more power than traditional training and to do it with a lower metabolic cost.5 It has also been reported that this type of training favors neural conduction and contributes to the prevention and improvement of health
  Interventions: Other: Group B. Eccentric exercises training

INTERVENTIONS:
Other: Group A Funtional massage therapy and eccentric exercise in lower limb — Functional Massage (FM) on lower limb. FM is a therapeutic technique that incorporates joint motion with massage to treat musculotendinous pain and impairments. Eccentric exercises training for lower limb. It can be useful in strengthening the muscles of the lower limbs, and promoting gait performance.
  Arms: Group A Functional massage in addition to eccentric exercise in paretic lower limb
Other: Group B. Eccentric exercises training — Eccentric exercises training and therapeutic exercise is a type of physical activity used to treat or prevent injuries and improve functional outcomes. Eccentric exercises focuses on movements, or phases of a movement, that lengthen the muscles. Some examples of eccentric exercise include lowering into a squat or lowering into a press-up. In contrast, when a person pushes out of a squat or press-up, this shortens the muscles. This is known as concentric movement
  Arms: Group B Eccentric exercise in paretic lower limb

SUMMARY:
Stroke is currently the leading cause of mortality in women, the second in men and the leading cause of disability in older adults. One of the most challenging sequelae after stroke is increased muscle tone due to spasticity, which alters muscle function. Functional massage therapy focuses on enhancing the function of muscles, joints, and connective tissues to improve movement and reduce pain. On the other hand, eccentric exercise, aids in the recovery of physical functions and is effective in managing spasticity improving muscle coordination and flexibility. It is essential to underline that the strength of evidence regarding these effects is considerable, supporting the implementation of these exercises in post-stroke treatment. In this context, an intervention combining functional massage with eccentric exercise on the lower limb is proposed for stroke survivors in the chronic phase. The goal of this crossover study is to analyze the effects of functional massage combined with eccentric exercise versus eccentric exercise alone on the effects of muscle tone, due to spasticity, of the lower limb in patients with chronic stroke. The Secondary Objectives are to analyze the effects of functional massage combined with eccentric exercise versus eccentric exercise alone on the improvement of ROM of the hip, knee and ankle joints, gait speed, lower limb function, quality of life and reduction of stress, anxiety and depression in patients with chronic stroke. The number of patients to be treated will be 8, the numbers of visits per patient will be 8 at the facilities of the university. Functional massage is a manual therapy technique that combines rhythmic passive mobilization of the joint, together with compression and decompression of the musculature to be treated. Eccentric exercises on lower limb focuses on movements, or phases of a movement, that lengthen the muscles. Some examples of eccentric exercise include lowering into a squat or lowering into a press-up. However, there are few previous studies combining these approaches to reduce spasticity and muscle tone and improve functionality in post-stroke patients. Participation in this study carries minimal risk, which could include events such as ankle endorses or falls during gait speed assessment or during therapeutic exercise. To mitigate these risks, participants will be allowed to use assistive devices such as splints, ankle braces, canes, or crutches during the activities selected for intervention. Importantly, patients in the chronic phase of stroke, and not in the acute phase, are included due to the stability of their condition which allows for safer and more effective participation in the study.

DETAILED DESCRIPTION:
According to the WHO, stroke is the second leading cause of death and the third leading cause of disability globally, with an increasing trend in both low- and middle-income countries. The estimated global cost of stroke has exceeded US$721 billion, representing 0.66% of the world's Gross Domestic Product (GDP) (1). Between 1990 and 2019, there was a substantial increase in the stroke-related burden, with a 70.0% increase in stroke cases, a 43.0% increase in stroke-attributed deaths, a 102.0% increase in prevalent stroke cases, and a 143.0% increase in Disability-Adjusted Life Years (DALYs). It is noteworthy that the majority of this burden of stroke, with 86.0% of deaths and 89.0% of DALYs, is concentrated in Low Income Countries (LMICs) and Lower Middle Income Countries (LMICs).

Ischemic stroke represents the second leading cause of death worldwide, with a total of 5.9 million deaths. However, a decrease in mortality rates has been observed in women, young people and in regions with a high sociodemographic index. The highest Standardized Mortality Rates (SMRs) and DALYs associated with ischemic stroke have been observed for women, young people and regions with a high sociodemographic index ischemic stroke are mainly concentrated in Central Europe (2). In Spain, stroke ranks first as a specific cause of mortality in women and second in men, according to data from the National Institute of Statistics (INE) (3). It is also the leading cause of disability in individuals over 65 years of age. According to INE projections for 2022, it was estimated that more than 24,000 deaths would be related to cerebrovascular diseases.

deaths were estimated to be related to cerebrovascular diseases, with more deaths in women than in men. It is important to note that, despite the decrease in the number of deaths due to cerebrovascular diseases in the last decade, the number of deaths in women is higher than in men. The last decade, the Spanish population's knowledge of stroke is still deficient (4).

Spasticity, as one of the main sequelae after stroke, occurs in approximately 30% of patients (5) and gradually worsens over time in the absence of adequate treatment, producing changes in muscle tissue such as hypertonia. Hypertonia alters motor function. It is defined as body functions related to muscle force and endurance, control over and coordination of voluntary movements, and movement patterns associated with walking, running or other whole body movements.

Likewise, mental health disorders, such as depression, stress or anxiety, are among the leading causes of disability worldwide. The three most common mental health disorders after stroke are post-stroke depression, post-stroke anxiety and post-traumatic stress disorder (6). These disorders often go undetected after a stroke and can have a significant impact on mortality rates. Recent research has shown that mental health disorders after stroke are associated with decreased functional outcomes and reduced quality of life.

However, these disorders continue to be "under-diagnosed and under-treated". Stroke is a common challenge in all countries, and its incidence increases significantly with age. Quality of life assessment can serve both to understand stroke and to measure the effectiveness of post-event rehabilitation (7).

Primary Hypothesis Functional massage combined with eccentric exercise is more effective in reducing muscle tone, due to spasticity, of the lower extremity in patients with chronic phase stroke, compared to those who only perform therapeutic exercise.

Secondary Hypotheses Functional massage combined with eccentric exercise is more effective in improving the range of motion (ROM), gait speed, functionality of the lower extremity in patients in reducing stress, anxiety and depression and improving quality of life with chronic stroke compared to those who only perform eccentric exercise.

Primary Objective To analyze the effects of functional massage combined with eccentric exercise versus therapeutic exercise alone on the improvement of muscle tone, due to spasticity, of the lower extremity in patients with chronic stroke.

Secondary Objectives To analyze the effects of functional massage combined with eccentric exercise versus eccentric exercise alone on the improvement of joint range of motion (ROM) of the hip, knee and ankle joints, in increasing gait speed, on the improvement of lower extremity function, in the reduction of stress, anxiety and depression in improving the perception of quality of life in patients with chronic stroke.

Methods The study will be a crossover randomized controlled clinical trial composed of two groups, a group A (n = 4) and a group B (n = 4), single blind (assessor). The intervention will have a duration of 4 weeks per group, in total 8 weeks per participant. The randomization will serve to decide to which group each patient will be assigned, taking into account that this patient will then be assigned, after a bleaching period, to the other intervention. The participant will be assess at baseline (T0) postintervention (T1). Recruitment will take place in specialized neurological rehabilitation centers in the metropolitan area of Barcelona, Spain.

All evaluations and interventions will take place at the facilities of the Universitat Internacional de Catalunya (UIC), Sant Cugat campus.

The principal researcher of the study will be in charge of informing both the participants and the center about the details of the study, including: the recruitment method, inclusion and exclusion criteria for participation, objectives, duration, risks and benefits. Participants will be voluntarily recruited by registering for the study through a Google Forms form sent to the center.

Recruitment will start in April 2025 with an expected closure in June 2025. The number of recruits will start with 8 participants, for a pilot trial due to the current scarce scientific evidence and thus initiate a possible line of research with a greater recruitment of patients.

Prior to participation in the trial, the participant or his/her legal representative will obtain a copy of the informed consent, freely given, signed and dated. Once the consent has been signed, the principal investigator will perform an individualized evaluation of each participant to ensure their inclusion in the study, according to the previously established inclusion and exclusion criteria.

Method of assignment:

Participants will be assigned to group A (intervention) or group B (control) by means of a concealment system. The concealment of the sequence will be governed by a simple randomization procedure with random number generation by computer. The list generated by the allocation sequence will guarantee a security copy of this and will be delivered to the principal investigator in an opaque envelope, which will be stored under lock and key at the facilities of the Universitat Internacional de Catalunya (UIC), until the end of the allocation process. This measure will guarantee the concealment of the list and avoid any possible bias during the process. Once the process is completed, the principal investigator will be in charge of assigning the interventions to the participants.

Masking:

The study will be governed by a single-blind masking procedure. To avoid efficacy bias in the study results, masking will be performed only to the assessor and will not be blinded to participants or intervenors (physical therapists). In the event of the presence of a serious adverse event related to the health or safety of a participant, the principal investigator should document whether unblinding is permitted. In the event that unblinding or any modification or correction of data occurs, the principal investigator should include the date and initials on the document, without obscuring the original data.

It will be ensured that all information collected during the clinical trial is recorded, managed and archived in a manner that facilitates its accurate communication, interpretation and verification. In addition, the confidentiality of records that may identify the participants will be preserved, in accordance with the applicable legislative regulations and respecting their privacy. To this end, when the patient signs the informed consent form, he/she will be assigned a code that will keep his/her name anonymous.

Intervention procedure:

During the first assessment, participants' personal data, anthropometric data, assessment of lower extremity muscle tone using the Modified Ashworth Scale (MAS) and the MyotonPRO will be collected. The ROM of the hip, knee and foot joints will also be measured with an inclinometer; gait speed (4 meters); lower extremity motor function with the Fugy-Meyer Scale; level of depression, anxiety and stress with the Depression, Anxiety and Stress Scale (DASS-21) and quality of life with the EQ-5D-5L Scale. In addition, participants will be provided with a paper log to record their feelings, as well as any adversity experienced, both at the beginning and at the end of the intervention. This log will be collected and stored under lock and key by the evaluators at the end of each session.

Evaluators should have a valid degree in physiotherapy, be registered with the college of physiotherapists and have at least 5 years of experience in neurological rehabilitation.

Material The intervention will require a stretcher where the passive and active functional massage and the pre- and post-intervention assessments that require it will be performed; the MyotonPRO for the assessment of muscle tone; a chair without armrests and without wheels for the eccentric exercise; an inclinometer for assessing the range of motion (ROM) of the hip, knee and leg joints; a stopwatch for recording walking speed; a wedge with slight elevation and an anti-slip disk for active eccentric exercise of the lower limb; a wedge with slight elevation and an anti-slip disk for active eccentric exercise of the lower limb; and a chronometer for recording walking speed.

Description of the intervention The intervention will be developed in two phases: in the first phase, group A will receive the intervention, while, in the second phase, this same group will act as the control group. The interventions will be carried out during 4 weeks, 4 sessions per group, with a duration of 90 minutes per session for the intervention group and one session of 45 minutes for the control group. Each session will include eccentric exercise comprising three active eccentric lower limb exercises for all participants. In addition, the intervention group will receive the passive functional massage technique on the lower limb for 30 minutes, according to the patient's tolerance.

In the forth week, group B, initially acting as a control group, will begin to receive the full intervention, incorporating functional massage in addition to the usual eccentric exercise.

In case of illness, cognitive impairment, difficulty in concentration or anxiety during the intervention, the participant will have the option to leave the study at any time. In addition, he/she will be able to rejoin the study, as long as the break period does not exceed 2 weeks.

Data Analysis Evaluation of experimental and statistical results: the selection of the most appropriate statistical software is in progress. However, the intention is to employ a rigorous approach to data analysis, which will probably include the use of regression models. In these models, the study outcomes will be considered as the dependent variable and the intervention group (experimental or control) as the main independent variable. The possibility of including other independent variables through a systematic method of variable selection, such as that proposed by Hosmer and Lemeshow, will also be explored to ensure the robustness of our analyses.

The study variables will be recorded in two time periods: at the beginning of the intervention (T0) and at the end of the intervention, 4 weeks (T1) with the validated scales and instruments . The research team will instruct all physical therapists in the use of the measurement instruments, including the MyotonPro and inclinometer.

Method of assignment:

Participants will be assigned to group A (intervention) or group B (control) by means of a concealment system. The concealment of the sequence will be governed by a simple randomization procedure with random number generation by computer. The list generated by the allocation sequence will guarantee a security copy of this and will be delivered to the principal investigator in an opaque envelope, which will be stored under lock and key at the facilities of the Universitat Internacional de Catalunya (UIC), until the end of the allocation process. This measure will guarantee the concealment of the list and avoid any possible bias during the process. Once the process is completed, the principal investigator will be in charge of assigning the interventions to the participants.

Masking:

The study will be governed by a single-blind masking procedure. To avoid efficacy bias in the study results, masking will be performed only to the evaluator and will not be blinded to participants or interventors (physical therapists). In the event of the presence of a serious adverse event related to the health or safety of a participant, the principal investigator should document whether unblinding is permitted. In the event that unblinding or any modification or correction of data occurs, the principal investigator should include the date and initials on the document, without obscuring the original data.

It will be ensured that all information collected during the clinical trial is recorded, managed and archived in a manner that facilitates its accurate communication, interpretation and verification. In addition, the confidentiality of records that may identify the participants will be preserved, in accordance with the applicable legislative regulations and respecting their privacy. To this end, when the patient signs the informed consent form, he/she will be assigned a code that will keep his/her name anonymous.

Ethical considerations:

Prior to initiation of the trial, foreseeable risks and inconveniences shall be considered in relation to the expected benefit, both to the individual trial subject and to society. The trial should be initiated and continued only if the anticipated benefits justify the risks. The rights, safety, and welfare of the trial participants shall be the most important considerations and shall prevail over the interests of science and society.

The clinical trial will be conducted in accordance with the Declaration of Helsinki 2024 and guidelines for research involving human subjects. This study will receive approval from the Human Research Ethics Committee and will be registered in the ClinicalTrials.gov Registry.

All participants, including legal guardians, will receive direction from the principal investigator on all aspects of the trial, including written information and Clinical Research Ethics Committee (IRB) approval.

If they wish to participate in the study, they will voluntarily sign a written informed consent statement. Informed written European data protection consent (14) will also be obtained from participants or legal guardians for the publication of any potentially identifiable images or data included in the trial. Participants will be informed that they may leave the study at any time without affecting their usual care.

Impact of the study and expected results At the end of the intervention, significant changes in muscle tone and functionality of the affected lower extremity are expected to be observed in patients with chronic phase stroke who received functional massage and therapeutic exercise, compared to those who received only therapeutic exercise. This combination of massage and therapeutic exercise is designed to improve mobility and reduce increased muscle tone due to spasticity, potentially improving patients' perception of quality of life.

Improved Functionality and Mobility: A marked improvement in the reduction of increased muscle tone in the lower extremity is expected, which should be reflected in improved mobility and functionality in daily activities.

1. Reduction of associated symptoms and improvement of emotional well-being: Functional massage is expected to bring additional benefits in the reduction of associated symptoms such as pain and fatigue, as well as in emotional regulation, contributing to the reduction of depression, stress and anxiety. This could increase the patient's motivation and participation in the rehabilitation process.
2. Impact on perception of quality of life: With the combination of functional massage and eccentric exercise, we seek to substantially improve the quality of life of participants, providing a more comprehensive tool for the management of post-stroke sequelae.
3. Long-term outcome evaluation: In addition, follow-up evaluations are proposed to investigate the sustainability of the benefits observed with additional massage sessions and at different stages of stroke, such as the subacute phase, to better understand the temporality and duration of the effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes ≥ 18 years of age.
2. Adults who have been diagnosed with an ischemic or hemorrhagic stroke, according to the diagnostic criteria established by the WHO; corresponding to ICD-11 in January 2022, as confirmed by CT or MRI
3. Stroke ≥ 6 months
4. Hospital discharge
5. Stable condition
6. Ability to understand and follow simple instructions
7. Ability to read, write and speak Spanish or Catalan with acceptable visual and auditory acuity
8. Living in the Barcelona metropolitan area
9. Able to comply with scheduled visits, treatment plan, and other trial procedures
10. Increased muscle tone in Lower Extremities (EEII) according to the modified Ashworth Scale (MAS) grade ≥ 1+ <4 11) Voluntary activation capacity and muscle strength in Lower Extremities (EEII) according to Daniels Scale grade ≥ 3 12) Ability to walk 10 meters, without assistance from third parties. 13) Minimum grade of 7 in depression, 5 in anxiety and 10 in stress according to the Depression, Anxiety and Stress Scale (DASS-21).

Exclusion Criteria:

1. Nervous system disease and/or cardiac, pulmonary dysfunction/failure.
2. History of mental disorders and/or cognitive impairment that make it difficult or impossible to follow instructions ≤ 21 Folstein's Mini Mental Test (MMSE)
3. Hearing impairment
4. History of psychotropic drug use in the last 6 months
5. Consumption of drugs to reduce spasticity or having undergone botulinum toxin treatment in the last 3 months.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Muscle tone will be assessed by modified Ashworth scale and Myoton pro. | Baseline and posttreatment at 4 weeks and at 8 weeks
  Muscle tone (residual muscle tension or tonus) is the continuous and passive partial contraction of the muscles, or the muscle's resistance to passive stretch during resting state. It helps to maintain posture and declines during REM sleep.Muscle tone is regulated by the activity of the motor neurons and can be affected by various factors, including age, disease, and nerve damage as spasticity.
  Modified Ashworth scale is performed by extending the patients limb's first from a position of maximal flexion to maximal extension (the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion. 0 is no increase in tone and 4 limb rigid in flexion or extension. The Myoton recording of dynamic tissue response in the form of physical displacement and oscillation acceleration signal and the subsequent computation of parameters characterizing the State of Tension, Biomechanical and Viscoelastic properties.

SECONDARY OUTCOMES:
Range of Motion (ROM) of the hip, knee and foot joints will be assessed by inclinometer. | Baseline and posttreatment at 4 weeks and at 8 weeks
  Range of motion is the capability of a joint to go through its complete spectrum of movements. It can be passive or active. Passive range of motion can be defined as what is achieved when an outside force, such as a therapist, causes movement of a joint. It is usually the maximum range of motion.
Gait speed will be assessed by 4 meters walking test at confortable pace and maximum pace. | Baseline and posttreatment at 4 weeks and at 8 weeks
  Gait speed is a key parameter to be assessed as it has often been considered a sixth vital sign. Gait speed tests can be administered at a comfortable pace (self-selected) or a fast pace (maximum without running). Executing the test at two paces can provide a more complete picture of an individual than either pace alone. A comfortable pace is useful for identifying gait ability in a clinical setting, and a fast pace may reflect the individual's activity level in the community, performing activities such as traversing pedestrian crossings. A rapid decline in gait speed is associated with an increased mortality risk. In addition, gait speed indicates whether the patient can ambulate in the community with a certain degree of safety, and it can be associated with motor function and functional mobility imbalance, and quality of life. Importantly, the literature has shown that the gait speed differs between sexes in the elderly.
Functionality of lower limb will be assessed by 30 seconds sit-to-stand and lower limb Fugl meyer scale | Baseline and posttreatment at 4 weeks and at 8 weeks
  The functionality of lower limb is to provide stability and support to the rest of the body, and through articulations with the femur and foot/ankle and the muscles attached to these bones, provide mobility and the ability to ambulate in an upright position.
Self-perceived emotional burden like stress, anxiety and depression will be assessed by Depression, Anxiety and Stress Scale-21 (DASS-21) | Baseline and posttreatment at 4 weeks and at 8 weeks
  Exposure to acute and chronic stress has a broad range of structural effects on the brain. The brain areas commonly targeted in the stress response models include the hippocampus, the amygdala, and the prefrontal cortex. Studies in patients suffering from the so-called stress-related disorders -embracing post-traumatic stress, major depressive and anxiety disorders in stroke survivors. DASS-21 is a Questionnaire short version (21 item) of a 42-item self report instrument designed to measure three related negative emotional states: depression, anxiety and tension/stress. The rating scale is as follows:
  0 Did not apply to me at all, Applied to me to some degree, or some of the time, 2 Applied to me to a considerable degree or a good part of time and 3 Applied to me very much or most of the time.
Quality of life and health status will be assessed by EuroQoL-5D-5L. | Baseline and posttreatment at 4 weeks and at 8 weeks
  Quality of life (QoL) is a concept which aims to capture the well-being, whether of a population or individual, regarding both positive and negative elements within the entirety of their existence at a specific point in time.
  Health status is a measure of how people perceive their health. Reported health status is a predictor of important health outcomes including mortality, morbidity, and functional status. Health is a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity. The enjoyment of the highest attainable standard of health is one of the fundamental rights of every human.
  EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ramón Rodríguez Rubio Pere Ramón Rodríguez-Rubio, PhD, Study Director — Universitat Internacional de Catalunya; Pere Ramón Rodríguez-Rubio Rodríguez-Rubio, PhD, Study Chair — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat Del Vallés, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Rueda L, Cabanas-Valdes R, Salgueiro C, Perez-Bellmunt A, Rodriguez-Sanz J, Lopez-de-Celis C. Immediate effects of TECAR therapy on lower limb to decrease hypertonia in chronic stroke survivors: a randomized controlled trial. Disabil Rehabil. 2025 Mar;47(5):1214-1223. doi: 10.1080/09638288.2024.2365992. Epub 2024 Jul 3. PMID 38958103
- [Background] Garcia-Rueda L, Cabanas-Valdes R, Salgueiro C, Rodriguez-Sanz J, Perez-Bellmunt A, Lopez-de-Celis C. Immediate Effects of TECAR Therapy on Gastrocnemius and Quadriceps Muscles with Spastic Hypertonia in Chronic Stroke Survivors: A Randomized Controlled Trial. Biomedicines. 2023 Nov 4;11(11):2973. doi: 10.3390/biomedicines11112973. PMID 38001972
- [Background] Fan J, Li X, Yu X, Liu Z, Jiang Y, Fang Y, Zong M, Suo C, Man Q, Xiong L. Global Burden, Risk Factor Analysis, and Prediction Study of Ischemic Stroke, 1990-2030. Neurology. 2023 Jul 11;101(2):e137-e150. doi: 10.1212/WNL.0000000000207387. Epub 2023 May 17. PMID 37197995
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Cabanas-Valdes R, Calvo-Sanz J, Serra-Llobet P, Alcoba-Kait J, Gonzalez-Rueda V, Rodriguez-Rubio PR. The Effectiveness of Massage Therapy for Improving Sequelae in Post-Stroke Survivors. A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Apr 21;18(9):4424. doi: 10.3390/ijerph18094424. PMID 33919371
- [Background] Cabanas-Valdes R, Garcia-Rueda L, Salgueiro C, Perez-Bellmunt A, Rodriguez-Sanz J, Lopez-de-Celis C. Assessment of the 4-meter walk test test-retest reliability and concurrent validity and its correlation with the five sit-to-stand test in chronic ambulatory stroke survivors. Gait Posture. 2023 Mar;101:8-13. doi: 10.1016/j.gaitpost.2023.01.014. Epub 2023 Jan 20. PMID 36696822
- [Background] Plasencia RR, VAN Zant J, Charron SC, Manderachia NM, Dickson J, Malek MH. Massage prior to exercise delays the onset of the physical working capacity at the fatigue threshold (PWCFT). J Sports Med Phys Fitness. 2025 May;65(5):650-656. doi: 10.23736/S0022-4707.24.16288-3. Epub 2024 Nov 11. PMID 39526873
- [Background] Clos P, Lepers R, Garnier YM. Locomotor activities as a way of inducing neuroplasticity: insights from conventional approaches and perspectives on eccentric exercises. Eur J Appl Physiol. 2021 Mar;121(3):697-706. doi: 10.1007/s00421-020-04575-3. Epub 2021 Jan 2. PMID 33389143
- [Background] Kinoshita Y, Osawa G, Morita T, Kawauchi M, Minowa T. [Diabetic glomerular sclerosis]. Nihon Rinsho. 1969 Aug;27(8):2045-53. No abstract available. Japanese. PMID 5390411
- [Background] Kwakkel G, Stinear C, Essers B, Munoz-Novoa M, Branscheidt M, Cabanas-Valdes R, Lakicevic S, Lampropoulou S, Luft AR, Marque P, Moore SA, Solomon JM, Swinnen E, Turolla A, Alt Murphy M, Verheyden G. Motor rehabilitation after stroke: European Stroke Organisation (ESO) consensus-based definition and guiding framework. Eur Stroke J. 2023 Dec;8(4):880-894. doi: 10.1177/23969873231191304. Epub 2023 Aug 7. PMID 37548025
- See also: Functional massage therapy focuses on enhancing the function of muscles, joints, and connective tissues to improve movement and reduce pain. Unlike general massage techniques aimed at relaxation, this method is goal-oriented and highly targeted. — https://www.spatheory.com/spa-theory-wellness-beauty-blog/functional-massage-therapy
- See also: Eccentric exercise focuses on movements that lengthenTrusted Source the muscles. For example, when someone lowers into a squat, their leg muscles lengthen. Eccentric movements require less oxygen and energy than other types of movement. — https://www.medicalnewstoday.com/articles/eccentric-exercise
- See also: The Hospital morbidity survey provides information on hospital discharges with hospitalisation based on the main diagnosis associated with the discharge. The main objective is to know the demographic and health characteristics of patients in Spain. — https://www.ine.es/dyngs/INEbase/en/operacion.htm?c=Estadistica_C&cid=1254736176778&menu=ultiDatos&idp=1254735573175